CLINICAL TRIAL: NCT02367443
Title: Hypofractionated Accelerated Radiotherapy With Concomitant Full Dose Chemotherapy for Locally Advanced Non-Small Cell Lung Cancer: Phase I/II Study
Brief Title: Hypofractionated Accelerated Radiotherapy With Concomitant Chemotherapy for NSCLC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Independent Public Care Health Facility of the Ministry of the Interior and Warmian & Mazurian Oncology Centre (Other)
Responsible Party: Principal Investigator, Lucyna Kepka, Prof., Independent Public Care Health Facility of the Ministry of the Interior and Warmian & Mazurian Oncology Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CentralHMIA
Record Dates: First submitted 2015-02-12; First posted 2015-02-20 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: radiotherapy; therapeutic use; Radiation; non-small cell lung cancer; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- one group (Experimental): Radiation: Hypofractionated accelerated Radiotherapy with concomitant full dose Chemotherapy
  Interventions: Radiation: Radiation

INTERVENTIONS:
Radiation: Radiation — Radiation: Accelerated Hypofractionated radiotherapy with full dose Chemotherapy

SUMMARY:
This is a phase I/II trial on concomitant RT-full dose CHT using accelerated hypofractionation schedule as currently being in routine use in Poland for sequential combination or RT alone. Objectives of the study are: to estimate rate of grade ≥ 3 CTCAE adverse effects related to treatment and to estimate tumor control, progression free-survival, and overall survival in patients treated with this regimen. Stage III NSCLC patients are treated according to the following schedule: RT: 58.8 Gy in 21 fractions (2.8 Gy/fraction, 5 times a week, 6 times in the third week; CHT concomitant with RT (2 cycle of Cisplatinum and Vinorelbine, every 21 days). Feasibility of the studied approach is evaluated by scoring the toxicity during RT-CHT and therafter, as well as percentage of treatment completion; efficacity is evaluated by estimation of local control and survival. If toxicity and efficacity are similar or better than those observed in modern series of conventionally fractionated RT-CHT, the studied regimen will become a routine treatment schedule in our institution in order to spare RT resources. In the future, a randomized comparison of the studied schedule with conventionally fractionated RT-CHT for locally advanced NSCLC is also planned.

DETAILED DESCRIPTION:
1. Background Lung cancer is the most common malignancy in Poland. In 2013, the annual lung cancer incidence in Poland was 175/100 000 in men and 95/100 000 in women, substantially higher than the EU value. Poland and UK are the first countries in Europe, where the mortality from lung cancer has overtaken the mortality from breast cancer and became the first cause of mortality from cancer in women. Thus besides the problem of prevention, the efficient and rational from economical point of view treatment of lung cancer is one of the crucial problems in Polish healthcare system. Prolongation of overall treatment time is deleterious for patients with locally advanced (LA) - non-small cell lung cancer (NSCLC) even if radio-chemotherapy (RT-CHT) is used. Current standard of treatment for LA-NSCLC is concurrent radio-chemotherapy (RT-CHT), because survival benefit with the increase of esophageal toxicity was demonstrated in a meta-analysis. Acceleration of radiotherapy (RT) via hyperfractionation results in survival benefit as it was shown also in a meta-analysis but at the expense of higher esophageal toxicity Hyperfractionated RT schedules were used with low-doses of CHT, because of the fear of accumulation of acute toxicity Hyperfractionation represents an additional burden for equipment, staff and health care system and cannot be routinely realized, especially in limited .resources setting. For patient, it is also associated with higher treatment cost, i.e. by payment of cost of transport twice a day.

   Alternative for acceleration of RT time is the use of hypofractionated RT schedule. Such a radiation schedule is in the routine use in some countries. However, hypofractionation has been often considered as palliative approach and even in limited resources countries is still rarely proposed for curatively treated patients. In only three out of 36 (8%) analysed Eastern and Central European centres that responded in the IAEA pattern of care survey, the hypofractionation was used for curative treatment of LA-NSCLC. We have also very few data from prospective studies that report on the concomitant hypofractionated RTwith full dose CHT. The RTOG 0117 study arm that used slightly hypofractionated RT schedule with dose escalation (75.25 Gy with 2.15 Gy fractional dose) and concomitant full-dose CHT was interrupted because of the excessive toxicity. However, the total dose escalation used in this study might be a reason for a failure of such an approach. Recently, the concept of dose escalation with concomitant CHT has been compromised for LA-NSCLC. When using hypofractionation, the total radiation dose should probably be adapted to correspond to biological doses of around 66 Gy, because we have reports that confrm safety of such a schedule. In opposite to that the dose escalation using hypofractionation for central tumors led to the excessive long-term toxicity due to the bronchial tree stenosis and perforations. In a few centers in Poland, the hypofractionated RT with total dose of 58.8 Gy in 21 fractions (in 4 weeks; in the third week 6 fractions are given) following two cycles of CHT or as RT alone is routinely used. Safety and efficacy of this approach was established in a phase II prospective trial. A question arises if such a RT schedule may be used concurrently with CHT. Given the proven benefit of concurrent RT-(full dose)CHT in stage III NSCLC, data on the value of overall treatment time and in order to spare RT resources we have decided to conduct a phase I/II trial on concomitant RT-(full dose)CHT using accelerated hypofractionation schedule as currently being in routine use in Poland for sequential combination or RT alone. Confirmation that toxicity and outcome in terms of local control and overall survival are similar to those observed in contemporary series of conventionally fractionated RT-CHT will lead to the incorporation of this schedule into routine practice in Poland. Such a schedule with shortened overall treatment time via hypofractionation will contribute to essential sparing of RT resources, still insufficient in Poland. Positive outcome of this study may be also a basis for future conduction of phase III study that compares conventionally fractionated RT-CHT with accelearated hypofractionated RT-CHT for stage III NSCLC.
2. Objectives of the study:

   To estimate toxicity and efficacy of accelerated hypofractionated RT combined with concurrent full-dose CHT for locally advanced NSCLC.

   STUDY HYPOTHESIS:

   RTOG/EORTC grade III and higher esophageal or pulmonary acute toxicity will not be higher than in conventionally fractionated concurrent RT-CHT i.e. 25%.

   And Two-year overall survival rate will be at least 40% and median overall survival will be higher than 20 months.

   2.1. Main endpoints: A. To estimate rate of RTOG/EORTC grade III and higher esophageal and pulmonary toxicity and grade IV and higher CTCAE version 3.0 hematological toxicity within 6 months from start of treatment.

   B. To estimate overall survival two years after start of RT-CHT.

   2.2. Secondary endpoints: A. Rate of two-year local control. B. All types of toxicity (esophagus, lung, skin, kidney, heart) within two years after start of RT-CHT.

   C. Feasibility of the study (percentage of completion of both planned cycles of CHT and full dose of planned CHT delivery; completion of planned RT, breaks in treatment and prolongation of overall treatment time).
3. Inclusion criteria:

   * Pathological or cytological confirmation of the diagnosis of NSCLC
   * Confirmation of clinical stage III based on: clinical examination, CT of the chest and abdomen (PET-CT highly recommended), bronchoscopy, CT or MRI of the brain if suspicion of brain metastases
   * No abnormalities in blood count precluding administration of full doses of Cisplatin and Vinorelbine (Neutrophils ≥1.5x109/L; Platelets ≥100 x109/L; Hemoglobin >11 g/dl)
   * No abnormalities in renal and hepatic function precluding administration of full doses of Cisplatin and Vinorelbine (creatinine clearance >50 ml/minute, aminotransferases < 1.5 of upper limit of normal value)
   * Age <75
   * KPS: 80-100
   * FEV1 > 1 liter (except cases with very low body surface, when FEV1 should be >40%)
   * No chronic diseases causing contraindication to the use of CHT
   * No previous RT on the thoracic region
   * Informed consent of patient for the participation in the study
4. Exclusion criteria:

   * Lack of meeting all inclusion criteria
   * Presence of clinically examined supraclavicular lymph nodes
   * Malignant pleural or pericardial effusion
5. Schema of the study:

   Stage III NSCLC patients who met inclusion criteria and signed informed consent are treated according to following schedule:
   * RT: 58.8 Gy in 21 fractions (2.8 Gy/fraction, 5 times a week, 6 times in the third week [treatment on Saturday])
   * Two cycles of CHT concomitant with RT: D1 - Cisplatin i.v. 80 mg/m2, Vinorelbine 25 mg/m2 i.v.; D8 - Vinorelbine 25 mg/m2 i.v.; D22 - Cisplatin 80 mg/m2 i.v.; Vinorelbine 25 mg/m2 i.v.; D29 - Vinorelbine 25 mg/m2 i.v.

   Patients are followed once a week during RT-CHT for evaluation of toxicity, then one month after treatment completion and every three months up two years after treatment, every six months thereafter. CT of the chest is performed during f/up at every visit. Blood tests for hematological toxicity will be performed at least once a week during radiotherapy and at each follow-up visit thereafter. Other examinations will depend on the clinical needs.
6. Chemotherapy (CHT) 6.1. General rules: Two cycles of CHT (Cisplatin & Vinorelbine) will be administered during RT every 21 days.

   6.2. Antiemetics: All patients will receive antiemesis prophylaxis before and during administration of CHT. This prophylaxis is mandatory sixty minutes before Cisplatin infusion.

   Recommended drugs are: Dexamethasone (12 mg p.o. or i.v. D1 and 22; 8 mg p.o. or i.v. D2, D3, D4; D23, D24, D25); 5-HT3 receptor antagonists, f.ex. Ondansetron 8 mg. i.v. D1, D22; NK-1 receptor antagonists, f.ex. Aprepitant 125 mg p.o. D1, D22 and 80 mg D2, D3, D23, and D24.

   The use of all other and additional antiemetics and combinations are possible, depending on the clinical indications and individual tolerance of drugs. Routine premedication before administration of Vinorelbine is not required.

   6.3. Doses of CHT and their modifications 6.3.1. Dose of Cisplatin is calculated based on the body-surface area - 80 mg/m2; diluted in 1000 ml of sodium chloride 0.9% and given over two-hours in i.v. infusion D1 and D22; Cisplatin will be administered after i.v. injection of Vinorelbine.

   6.3.2. Dose of Vinorelbine is calculated based on the body-surface area - 25 mg/m2; diluted in 125 ml of sodium chloride 0.9% and given over 20 minutes in i.v. infusion D1, D8, D22 and D29.

   6.3.3. Doses of CHT will be modified in consecutive cycles depending of hematological toxicity. Neutrophils level before each cycle of CHT should be ≥1.5x109/L and platelets level should be ≥100 x109/L. In case of incidence of hematological toxicity, the drug doses will be modified according to the schema presented in Table 1.

   Table 1. CHT dose modifications for 2nd cycle of CHT depending on hematological toxicity observed at the first CHT cycle.

   Nadir of Platelets (x109/L) Nadir of Neutrophils (x109/L) Dose modification; Action taken >100 and > 1.5 100% 75-100 or 1.0-1.5 One week deferral <75 or <1.0 One week deferral and reduction of dose to 75% of initial dosing

   Persistent Grade III or higher CTC toxicity up to end of RT Persistent Grade III or higher CTC toxicity up to end of RT Discontinuation of Chemotherapy

   6.3.4. Hematopoietic growth factors won't be used for primary prophylaxis of febrile neutropenia.
7. Radiotherapy (RT)

   7.1. Target volume definition: Whole treatment will be planned in the three-dimensional (3D) planning system, according to the requirement of ICRU recommendations of planning, delivering and reporting doses of 3D-conformal radiotherapy (3D-CRT) [13]. IMRT technique won't be used for planning in this study.

   GTV will be considered as radiologically and bronchoscopically visualized tumor, as well as pathological regional lymph nodes (LN). Mediastinal and hilar LN will be considered as pathological if FDG-avid in PET-CT scan. In case of absence of abnormal FDG-uptake all LN with short axis diameter ≥1.5 cm will be considered as pathological and included in the GTV, unless clinical and radiological judgment will indicate with high probability other than malignant etiology of lymph node enlargement. Pathological confirmation of abnormal FDG up-take in regional lymph nodes won't be mandatory. In rare cases of lack of PET-CT for staging, LN with short axis diameter >1 cm will be considered as pathological, unless the formal exclusion of their metastatic origin is provided by radiologist, i.e. benign appearance.

   CTV: will be created by adding 0.5 cm to the GTV of primary tumor. Nodal CTV will consist of the whole LN station (LNS), in which pathological LN are found. Borders of LNS will be designed according to the guidelines of Michigan Atlas [14] with modification of Kepka et al. [15] for hilar motion uncertainty.

   PTV: will be created by adding 1 cm margin to the CTV. Sometimes PTV margin will be modified individually depending of respiratory motion and spirometry test's results of the patient.

   7.1. Radiotherapy planning: CT for planning will be done in therapeutic patient's position and immobilization as for all other thoracic localizations in the department. Scan thickness is 3 mm. The i.v. contrast use for planning is not mandatory.

   Dose will be prescribed in ICRU point; energy of 6 (or exceptionally 15) MV photons will be used.

   Dose per fraction: 2.8 Gy, RT once a day, 5 times a week in 1st, 2nd and 4th week of RT; 6 times a week in the 3rd week of RT (treatment on Saturday).

   Total dose: 58.8 Gy Dose homogeneity criteria: 95-107% of the prescribed dose; minimum dose of 90% will be also allowed in the PTV (as point dose).

   Doses for critical structures:

   Spinal cord: maximum dose - 45 Gy; 40 Gy for a length < 5 cm. Lung: mean dose ≤20 Gy (or less depending on individual physician decision if respiratory reserve of patient is limited); 35% of total lung volume receives ≤20 Gy Heart: 50% of heart volume receives less than 40 Gy; avoidance of hot-spot within this organ Esophagus: recommended mean dose <34 Gy; avoidance of hot-spots within this organ.

   7.2. Radiotherapy delivery: Physician will be present at the first RT session. The set-up verification with KV portals will be done and portal imaging for all therapeutic portals will be done and fused with respective DRR at the first RT session. MV cone beam verification will be possible at the request of the physician, but not mandatory. Next KV set-up verification will be realized at least once a weak. On-line and off-line QA procedures won't differ from those for other curative treatments in the RT Department.
8. Toxicity evaluation Early lung and esophageal toxicity will be scored according to the RTOG/EORTC scale once a week during radiotherapy, next one month after completion of RT, and in the third and sixth month after treatment. During the same follow-up visit all types of toxicity from other organs, like skin, heart will be scored according to the same scale [15].

   Late radiation toxicity will be evaluated after 6 months of follow-up every three months within two years and every six months thereafter according to the RTOG/EORTC scale.

   Hematological toxicity will be evaluated according to the CTCAE vs 3.0 [17] in the same intervals than esophageal and pulmonary toxicity during radiotherapy and thereafter, or more often if clinically indicated. Other types of CHT toxicity will be also reported according to the CTCAE scale, if they occur.
9. Evaluation of the outcome of RT-CHT CT of the chest will be done one month after treatment completion. Then CT of the chest as well as the physical examination and blood tests will be done at each follow-up visit. Other radiological examinations will be prescribed if clinically indicated.

   Overall survival will be estimated according to the Kaplan-Meier method and calculated from the first day of RT-CHT. Actual risk of loco-regional failure will also be estimated using the Kaplan-Meier method. Distant metastases occurrence and their sites will be scored and reported.
10. Number of patients and study duration Study will be conducted in one institution. Ethic Committee agreement for study conduction is required. It is planned to include 100 patients during first three years; minimum follow-up required after inclusion of last patient is one year. Thus planned time of study conduction is four years, meant as the time to the submission of publication that reports the outcome. Before that, the publication of interim analyses is allowed if judged as clinically and scientifically relevant by the investigators.
11. Predefined rules of study earlier halting or termination

    Study will be earlier terminated or appropriately modified after Investigators Meeting and consultation of Ethical Committee if:
    * After completion of 6 months of follow-up for first 10 included patients, the CTCAE hematological toxicity of grade IV or higher will occur in 3 or more patients and/or the grade III or higher RTOG/EORTC pulmonary or esophageal toxicity will occur in 3 or more patients, and also if two or more toxic deaths* will be reported.
    * After completion of 6 months of follow-up for first 30 included patients, the CTCAE hematological toxicity of grade IV or higher will occur in ≥30% of patients and/or the grade III or higher RTOG/EORTC pulmonary or esophageal toxicity will occur in ≥30% of patients, and also if three or more toxic deaths* will be reported.

      * Every toxic death will lead to the extra meeting of the study investigators in order to ascertain if immediate study modification is not necessary. Every death scored as for unknown reason will require an undertaking of all necessary steps to find all its circumstances to qualify with the highest possible probability its cause.
12. Expected outcomes of the study We expect to confirm prospectively the safety and efficacy of studied approach, meant as esophageal and pulmonary toxicity not higher and overall survival not lower than that observed in contemporary series with conventionally fractionated concurrent RT-CHT. After confirmation of the study hypothesis, a phase III study that compares the studied schedule with conventionally fractionated RT-CHT will be justified. The studied accelerated hypofractionated RT-CHT schedule may become routine treatment protocol for stage III NSCLC patients what will reduce treatment cost and enable better sparing of accessible RT technological resources.

ELIGIBILITY:
Inclusion Criteria:

* • Pathological or cytological confirmation of the diagnosis of NSCLC

  * Confirmation of clinical stage III based on: clinical examination, CT of the chest and abdomen (PET-CT highly recommended), bronchoscopy, CT or MRI of the brain if suspicion of brain metastases
  * No abnormalities in blood count precluding administration of full doses of Cisplatin and Vinorelbine (Neutrophils ≥1.5x109/L; Platelets ≥100 x109/L; Hemoglobin >11 g/dl)
  * No abnormalities in renal and hepatic function precluding administration of full doses of Cisplatin and Vinorelbine (creatinine clearance >50 ml/minute, aminotransferases < 1.5 of upper limit of normal value)
  * Age <75
  * KPS: 80-100
  * FEV1 > 1 liter (except cases with very low body surface, when FEV1 should be >40%)
  * No chronic diseases causing contraindication to the use of CHT
  * No previous RT on the thoracic region
  * Informed consent of patient for the participation in the study

Exclusion Criteria:

* Lack of meeting all inclusion criteria
* Presence of clinically examined supraclavicular lymph nodes
* Malignant pleural or pericardial effusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2014-03; Primary Completion 2019-10 (Actual); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Toxicity | 3 years
  Grade III and higher

SECONDARY OUTCOMES:
Survival | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Independent Public Health Care Facility and Warmian & Mazurian Oncology Centre, Olsztyn, Poland